CLINICAL TRIAL: NCT07170878
Title: Effect of Blueberry Supplementation on Liver Enzymes, Muscle Injury and Respiratory Parameter in Football Athletes: A Eight-Week Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, ASSOC. PROF., Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-95674917-108.99-164965
Record Dates: First submitted 2025-03-04; First posted 2025-09-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Performance
Keywords: Respiratory Parameter; Liver Enzymes; Muscle Damage; Blueberry; Football

STUDY DESIGN:
Intervention Model Description: Participants visited the laboratory 3 times. At the first visit, information about the study was given and try tests of the tests and training to be used were carried out. At the second visit, measurements of respiratory function and respiratory muscle strength and blood samples were taken. At the final visit, after 8 weeks of training, the measurements taken at the second visit were repeated.
  Eight Weeks Reinforcement Period Blueberry powder supplementation (26 g or ~1 cup fresh blueberry equivalent per day) was provided in 25 vacuum-sealed packets consisting of low bush wild blueberries (Vaccinium angustifolium Ait) sourced from Allen's Blueberries (Ellsworth, ME) and freeze-dried by Future Ceuticals (Momence, IL). Study participants consumed blueberry powders mixed with water, fruit juice, yoghurt or other products in the first meal of the day before each workout for 8 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supplementation Group (EG) (Experimental): group given blueberry supplement in addition to soccer training
  Interventions: Dietary Supplement: Blueberry Supplementation; Dietary Supplement: Supplementation Group
- CONTROL (No Intervention): The research group (Control Group (CG) (n:12): soccer training group;
- Reinforcement+Exercise (SEG) (Active Comparator): Reinforcement+Exercise (SEG) (n:12): the group who was given additional blueberry supplement in soccer training and 20 minutes of resistance band exercise)
  Interventions: Dietary Supplement: Blueberry Supplementation; Dietary Supplement: Supplementation Group

INTERVENTIONS:
Dietary Supplement: Blueberry Supplementation — The research group (Control Group (CG) (n:12): soccer training group; Supplementation Group (EG) (n:12): group given blueberry supplement in addition to soccer training; Reinforcement+Exercise (SEG) (n:12): the group who was given additional blueberry supplement in soccer training and 20 minutes of resistance band exercise) consisted of 36 male athletes in the football branch and regularly participating.
  Arms: Reinforcement+Exercise (SEG); Supplementation Group (EG)
Dietary Supplement: Supplementation Group — Supplementation + Exercise
  Arms: Reinforcement+Exercise (SEG); Supplementation Group (EG)

SUMMARY:
Abstract Background and objective: Regular Exercise causes physiological changes in the body. As a result, its impact on liver enzymes and muscle injury is unknown. The purpose of this study was to look into the effect of blueberry supplement taken in addition to football training on athlete muscle injury, liver enzymes and respiratory parameter. Methods: The present study comprised 36 male football players who volunteered for the study. The participants were divided into three groups: a Control Group (CG) (n=12), which performed only football training; a Supplementation Group (EG) (n=12), which received blueberry supplementation in addition to football training; and a Supplementation + Exercise Group (SEG) (n=12), which received blueberry supplementation and 20 minutes of exercise in addition to football training. A eight-week training program was implemented to the athletes three days per week in our study. The athletes' blood was drawn twice before and after training. The athletes' markers of muscle injury and liver enzymes were measured as a result of blood samples taken. The SPSS package program was used to examine the study's data.

DETAILED DESCRIPTION:
Original Research Effect of Blueberry Supplementation on Liver Enzymes, Muscle Injury and Respiratory Parameter in Football Athletes: A eight-Week Training Study Abstract Background and objective: Regular Exercise causes physiological changes in the body. As a result, its impact on liver enzymes and muscle injury is unknown. The purpose of this study was to look into the effect of blueberry supplement taken in addition to football training on athlete muscle injury, liver enzymes and respiratory parameter. Methods: The present study comprised 36 male football players who volunteered for the study. The participants were divided into three groups: a Control Group (CG) (n=12), which performed only football training; a Supplementation Group (EG) (n=12), which received blueberry supplementation in addition to football training; and a Supplementation + Exercise Group (SEG) (n=12), which received blueberry supplementation and 20 minutes of exercise in addition to football training. A eight-week training program was implemented to the athletes three days per week in our study. The athletes' blood was drawn twice before and after training. The athletes' markers of muscle injury and liver enzymes were measured as a result of blood samples taken. The SPSS package program was used to examine the study's data.

Keywords: Football, Blueberry, Muscle Damage, Liver Enzymes, Respiratory Parameter

1. Introduction Exercise is a type of physical activity that is done in leisure time to develop or maintain physical fitness, performance, or health. Exercise is recognized to have numerous beneficial impacts, including increased endurance, flexibility, strength, body shape maintenance, reduced risk of cardiovascular disease, and weight loss. The type, frequency, intensity, duration and progression of exercise should be regulated depending on individual factors. Since each individual's physical condition level, goals, health status and personal preferences are different, it is important to plan the exercise program individually. It can be challenging to provide a definitive answer without testing and receiving the person's physiological reactions concerning which sort of exercise will provide the most benefit, at what frequency, intensity, and duration.

   Muscle pain after exercise is thought to harm the muscles. Excessive stretching of the elastic and contractile tissues of the muscle during movement produces structural damage, which causes pain. The intensity, weight, and scope of the applied training all have an impact on the amount of damage that happens. Particularly in high-intensity training, oxidative stress is seen in the organism, followed by muscle damage in the organism, and finally, muscle pain occurs during and at the end of exercise as a reaction of neutrophils to inflammation. Creatine Kinase (CK) and Myoglobin creatine kinase (CKMB) are biochemical indicators that are used to detect muscle injury in an organism. Many enzymes are stored, secreted, and concentrated in the liver cells, which also act as a metabolic organ, and enzymes are released into the blood. The ALT (Alanine Amino transferase), AST (Aspartate Amino transferase), ALP (Alanine amino transferase) and LDH (Lactaid Dehydrogenase) enzymes released from these cells help determine whether there is any damage in the liver. Changes in liver enzyme values are noticed during heavy and rigorous exercise, and LDH, AST, and ALT enzymes are routinely utilized to detect hepatocellular injury. It is critical to minimize any muscle injury that may develop in the organism in order to ensure and maintain athletic performance.

   Otherwise, the hypertonicity of the respiratory muscles leading to their expansion results in a reduction in the movement of the spine, costal, and sternal regions. Disruptions in respiratory mechanics are often caused by the shortening of the respiratory muscle system. Factors contributing to this shortening include psychoneural factors (stress), muscle weakness, and inadequate physical activity. It is well known that long-term mechanical ventilation training can lead to oxidative stress and damage to the diaphragm. To assess muscle damage, CKMB and CK have been indicated as useful for evaluating inspiratory muscles.

   Blueberries are high in polyphenolic chemicals (most notably anthocyanins), which have antioxidant, anti-fatigue, and anti-inflammatory properties. Studies in the literature suggest that blueberry supplementation has the potential to provide various health benefits, including improving metabolic function, reducing inflammation and oxidative stress, enhancing vascular function, decreasing the risk of dementia, and promoting neuronal signaling. Additionally, there is evidence that the composition of the gut microbiome influences insulin receptor sensitivity and other aspects of metabolic and immune function, with these effects being partially mediated by increased cytokine expression. Specifically, the gut microbiota can be positively altered in response to dietary changes, including the consumption of bioactive compounds such as flavonoids. However, studies on the effects of blueberry supplementation on liver enzymes, muscle damage, and respiratory parameters are limited. The aim of this study is to investigate the effects of blueberry supplementation on liver enzymes, muscle injury, and respiratory parameters in football players.
2. Materials and Methods Study design and Participants This study was approved by the Ethics Committee of Elazığ University (2025/2; E-95674917-108.99-164965). Prior to the commencement of the study, participants were thoroughly informed about the study's content, purpose, and experimental design. Parents of those who agreed to participate signed an informed consent form. The inclusion criteria were as follows: (a) at least two years of active football experience, (b) age between 14 and 16 years, (c) good general health with no known respiratory or cardiovascular conditions, (d) provision of written informed consent, and (e) Playing football in Elazığspor. Exclusion criteria were as follows: (a) history of lung disease or current upper respiratory tract infections; (b) existing injury problems; (c) use of medications that could affect respiratory; (d) current smokers or individuals with a history of smoking within the past year; and (e) participation in similar studies within the last six months. A cross-sectional study was conducted, with the sample size determined using G*Power software. A power analysis (alpha = 0.05, power = 0.50, η2p = 0.8) showed that at least 10 participants were required for each group. In this study, the quota sampling method was employed to select a sample of thirty-six volunteer amateur football players with a minimum of two years of active working history in Elazığ province. The research group (Control Group (CG) (n:12): soccer training group; Supplementation Group (EG) (n:12): group given blueberry supplement in addition to soccer training; Reinforcement+Exercise (SEG) (n:12): the group who was given additional blueberry supplement in soccer training and 20 minutes of resistance band exercise) consisted of 36 male athletes in the football branch and regularly participating.

Participants visited the laboratory 3 times. At the first visit, information about the study was given and try tests of the tests and training to be used were carried out. At the second visit, measurements of respiratory function and respiratory muscle strength and blood samples were taken. At the final visit, after 8 weeks of training, the measurements taken at the second visit were repeated.

Pulmonary Function Tests (PFT) Peak expiratory flow (PEFmax ) and forced expiratory volume (FEV1), which is the volume that has been exhaled at the end of the first second of forced expiration), FEV1 / FVC (Tiffenau index), and After profound inspiration, the total exhaled volume forced vital capacity (FVC) were measured using an MGF Diagnostics CPFS/D USB spirometer. Each participant was fitted with a nose clip and instructed to take as deep a breath as possible through the mouth tube connected to the spirometer and blow as hard and fast as possible. Three trials were obtained and the largest of the three was selected for analysis. Artists with an FEV1 / FVC < 75% and those with a history of lung disease, upper respiratory tract infection, or current voice impairment were excluded. PFT was measured according to the 2002 guidelines of the American Thoracic Society and the European Respiratory Society (ATS/ERS). Subjects were verbally motivated to exert maximal effort in all respiratory tests.

Maximal Inspiratory (MIP) and Expiratory (MEP) Pressure Measurement MIP and MEP were measured using a portable hand-held mouth breathing pressure monitor (MicroRPM; CareFusion Micro Medical, Kent, UK) according to the 2002 guidelines of the American Thoracic Society and European Respiratory Society (ATS/ERS). After appropriate filters and holders were fixed, the nasal airway was closed using a clip. MIP measurements were started with residual volume and MEP measurements were started with total lung capacity. Measurements were repeated until a 5% difference between the two best findings was recorded as the mean cm H2O.

Training Program The research group was subjected to a four-week, ninety-minute football training regimen three days a week. 5-10 minutes of warm-up time, 50-60 minutes of football training, and 5-10 minutes of cool-down activities were completed as part of the program. Only the training program was used, with no blueberry given to the control group. Blueberry supplements were supplied to the supplement group, and a regular workout program was used. Stretching activities with resistance bands were done at the end of the training session by delivering blueberries to the supplement and exercise groups.

Warm-Up and Stretching (10 min.) Technical Training (20 min.) Physical Training (25 min.)

* 2 minutes of light jogging Dinamik Esneme
* High-knee walking (10 steps)
* Heel-to-butt walking (10 steps)
* Arm rotations (10 reps) Warming Up with the Ball
* Short dribbles and changes of direction with the ball at a slow pace. • Pass exchange between groups of 2 at a distance of 5-10 meters.
* Control and single pass, then control and pass.
* 1 touch (single ball) pass exchange • Slalom dribbling with cones (speed and control work).
* Shooting work after dribbling: Passing through cones and hitting a small target. • 10-meter sprint exercises (4 singles)
* Cross runs and sudden changes of direction (2 min.) Durability
* 3 sets of 1 minute light jogging + 30 seconds sprinting. Mini Match (15 Minutes)
* A 5v5 match on a small field or match that suits the number of players available.
* More ball control and playmaking oriented. Cool Down and Stretch (5 Minutes)
* Light-paced walking (2 minutes).
* Static stretching:
* Hamstring, quadriceps, calf and hip stretching exercises.
* Waist and shoulder stretching. Resistance Band Exercise 10-Minute Resistance Band Cool-Down Exercises

  1.Light Band-Assisted Stretching (3 minutes)
* Hamstring Stretch (1 minute) Sit on the floor with one leg extended and the band wrapped around your foot. Gently pull the band to stretch your hamstring. Hold for 30 seconds per leg.
* Quad Stretch (1 minute) Stand or lie on your side. Loop the band around your ankle and gently pull it towards your glutes. Hold for 30 seconds per leg.
* Calf Stretch (1 minute) Sit with one leg extended and wrap the band around the ball of your foot. Pull the band gently to stretch your calf. Hold for 30 seconds per leg.

  2. Shoulder and Arm Stretches (3 minutes)
* Overhead Tricep Stretch (1 minute) Hold the band behind your back with one hand reaching over your shoulder and the other behind your lower back. Gently pull to stretch your tricep and shoulder. Switch sides after 30 seconds.
* Chest Opener (1 minute) Hold the band behind your back with both hands and gently pull to open your chest. Hold for 30 seconds and repeat.
* Side Stretch (1 minute) Hold the band above your head with both hands. Gently pull the band as you lean to one side, stretching your obliques. Hold for 30 seconds per side.

  3. Lower Back and Hips (4 minutes)
* Seated Forward Fold (1 minute) Sit with your legs extended and the band around your feet. Pull yourself gently forward, feeling the stretch in your lower back and hamstrings. Hold for 1 minute.
* Hip Flexor Stretch (1 minute per side) Step into a lunge position and loop the band around your back leg's ankle. Pull gently while sinking into the stretch. Switch sides after 1 minute.
* Glute Stretch (1 minute) Lie on your back and place the band around one foot. Cross the opposite ankle over your knee, forming a figure-four shape. Gently pull on the band to stretch your glutes. Switch sides after 30 seconds.

Eight Weeks Reinforcement Period Blueberry powder supplementation (26 g or ~1 cup fresh blueberry equivalent per day) was provided in 25 vacuum-sealed packets consisting of low bush wild blueberries (Vaccinium angustifolium Ait) sourced from Allen's Blueberries (Ellsworth, ME) and freeze-dried by Future Ceuticals (Momence, IL). Study participants consumed blueberry powders mixed with water, fruit juice, yoghurt or other products in the first meal of the day before each workout for 8 weeks.

Nutrition Protocol Male footballers use energy availability (EA) > 25 kcal/kg fat-free mass (FFM) to maintain muscle mass during the competition period and avoid negative health consequences against lower levels of energy availability (Fagerberg, 2018). Meals during the day were taken at 3.5-hour intervals. The average daily calorie intake of the subjects was calculated as 2500--3500 kcal. A diet programme was prepared for footballers with 64.2% of calories coming from cho, 27.1% from protein and 8.7% from fat. The mean protein intake was 2.5 g/kg/day. Dietary intake of micronutrients was not adequate for the study subjects.

Collection and Analysis of Samples Blood samples were taken from the athletes in the research group twice, at the beginning and at the end of the exercise programme. ALT, AST, LDH, CK and CK-MB levels were determined as markers of muscle damage. Blood samples were taken from the athletes in sitting position and at rest. All examinations were analysed by professionals in a private medical laboratory using a Coulter Counter-S model (Coulter ®; STKS, Coulter Corp., Hialeah, FL, USA) from a 4 mL sample.

Statistical Analysis The SPSS statistical package tool was used to analyze the data. The data was normality tested and parametric tests were employed for the data that was found to be normally distributed. The "Paired Samples t" test was used for in-group comparisons, and the "One-way ANOVA" test was used for intergroup comparisons. Significance level was taken as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

a) at least two years of active football experience, (b) age between 14 and 18 years, (c) good general health with no known respiratory or cardiovascular conditions, (d) provision of written informed consent, and (e) Playing football in Elazığspor.

Exclusion Criteria:

1. history of lung disease or current upper respiratory tract infections;
2. existing injury problems;
3. use of medications that could affect respiratory;
4. current smokers or individuals with a history of smoking within the past year;
5. participation in similar studies within the last six months.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Change in muscle injury markers | 8 weeks
  Change in muscle injury markers (CK) from baseline to 8 weeks.
Change in liver enzyme levels | 8 weeks
  Change in liver enzyme levels (ALT) from baseline to 8 weeks.
Change in muscle injury markers | 8 weeks
  Change in muscle injury markers (CK-MB) from baseline to 8 weeks.
Change in liver enzyme levels | 8 weeks
  Change in liver enzyme levels (AST) from baseline to 8 weeks.
Change in liver enzyme levels | 8 weeks
  Change in liver enzyme levels (LDH) from baseline to 8 weeks.
Change in liver enzyme levels | 8 weeks
  Change in liver enzyme levels (ALP) from baseline to 8 weeks.

SECONDARY OUTCOMES:
Change in pulmonary function parameters | 8 weeks
  Change in pulmonary function parameters (FVC) after 8 weeks.
Change in maximal inspiratory pressure | 8 weeks.
  Change in maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).
Change in pulmonary function parameters | 8 weeks
  Change in pulmonary function parameters (FEV1) after 8 weeks.
Change in pulmonary function parameters | 8 weeks
  Change in pulmonary function parameters ( FEV1/FVC ) after 8 weeks.
Change in pulmonary function parameters | 8 weeks
  Change in pulmonary function parameters ( PEFmax) after 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane Univetsity, Gümüşhane, Kelkit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF